CLINICAL TRIAL: NCT04208958
Title: Phase 1 Study of VE800 and Nivolumab in Patients With Selected Types of Advanced or Metastatic Cancer
Brief Title: Study of VE800 and Nivolumab in Patients With Selected Types of Advanced or Metastatic Cancer
Acronym: ConsortiumIO
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Vedanta Biosciences, Inc. (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VE800-001
Record Dates: First submitted 2019-12-16; First posted 2019-12-23 (Actual); Results first posted 2023-08-29 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2023-03

CONDITIONS: Metastatic Cancer; Melanoma; Gastric Cancer; Gastroesophageal Junction Adenocarcinoma; Colorectal Cancer
Keywords: Metastatic Cancer; VE800; Nivolumab; Opdivo; Melanoma; Gastric Cancer; Gastroesophageal Junction Adenocarcinoma; GEJ Adenocarcinoma; Colorectal Cancer; CRC-MSS; Vedanta; BMS
MeSH Terms: conditions — Neoplasm Metastasis; Melanoma; Stomach Neoplasms; Colorectal Neoplasms | interventions — Nivolumab; Vancomycin

STUDY DESIGN:
Intervention Model Description: This study was designed to help determine the safety and effectiveness of the study drug, VE800, in combination with nivolumab in patients with advanced/metastatic cancer.
  The following cohorts of patients with advanced/metastatic cancer were enrolled:
  * Melanoma
  * Gastric/gastroesophageal junction (GEJ) adenocarcinoma
  * Colorectal cancer (microsatellite-stable) (CRC-MSS)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- VE800 combination treatment with nivolumab (Experimental): Subjects received 5 days of oral vancomycin, followed by daily VE800 in combination with nivolumab every 4 weeks.
  Interventions: Biological: VE800; Drug: Nivolumab; Drug: Vancomycin Oral Capsule

INTERVENTIONS:
Biological: VE800 — VE800 is an orally administered (PO) live biotherapeutic product (LBP) consisting of 11 distinct nonpathogenic, nontoxigenic, commensal bacterial strains manufactured under Good Manufacturing Practice (GMP) conditions. These strains were selected for their ability to induce an immune response.
Drug: Nivolumab — Nivolumab is an approved medication that blocks antibodies for certain types of cancer.
  Other Names: Opdivo
Drug: Vancomycin Oral Capsule — Vancomycin is an antibiotic used to treat or prevent infection.
  Other Names: Vancocin

SUMMARY:
This study evaluated the safety and efficacy of VE800 in combination with nivolumab in patients with selected types of advanced or metastatic cancer

DETAILED DESCRIPTION:
CONSORTIUM-IO was the first-in-human multicenter, open-label study; the main objectives were to evaluate:

* Safety and tolerability of VE800 in combination with nivolumab
* Efficacy as measured by objective response rate

The study planned to enroll approximately 111 patients with melanoma, gastric/gastroesophageal junction (GEJ) adenocarcinoma, or microsatellite-stable (MSS) colorectal cancer (CRC).

Nivolumab is already approved by the U.S. Food and Drug Administration (FDA), however, it is not approved for the study cancer indications. VE800 was the investigational product, which was designed to enhance the immune response to the tumor.

ELIGIBILITY:
Partial Inclusion Criteria:

* Patients with advanced or metastatic cancer who had received no more than 3 lines of prior systemic therapy for advanced/metastatic disease.
* Histologically diagnosed advanced (unresectable) or metastatic cancer with at least one measurable lesion as per RECIST 1.1
* Tumor lesions amenable for biopsy, if deemed safe by the investigator
* Toxicity from prior cancer therapy should have resolved to Common Terminology Criteria for Adverse Events (CTCAE) Grade ≤ 1 (excluding alopecia and neuropathy, where up to Grade 2 residual was allowed)

Partial Exclusion Criteria:

* Prior treatment with immune checkpoint inhibitor (iCPI) (Note: this criterion did not apply to patients with melanoma)
* Receipt of any conventional or investigational systemic anti-cancer therapy within 21 days prior to the first dose of vancomycin
* Concurrent chemotherapy, immunotherapy, biologic, or hormonal anti-cancer therapy. Agents such as bisphosphonates or denosumab were acceptable as prophylaxis for bone metastasis.
* Patients must not have received a transfusion (platelets or red blood cells) within 4 weeks of the first dose of study treatment
* Patients with an active, known or suspected autoimmune disease. Patients with type I diabetes mellitus, hypothyroidism only requiring hormone replacement, skin disorders (such as vitiligo, psoriasis, or alopecia) not requiring systemic treatment were permitted to enroll.
* Patients with known active hepatitis (e.g., hepatitis B or C) NOTE: Patients with previously treated hepatitis B or C were permitted to enroll if there was evidence of documented resolution of infection.
* Received a fecal transplant, spore or other preparation of fecal material, isolated bacterial products, genetically modified bacteria, or VE800

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2020-01-23 (Actual); Primary Completion 2021-08-26 (Actual); Study Completion 2023-02-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Judy Wang, MD, Principal Investigator — SCRI - Florida Cancer Specialists - Sarasota Cattlemen Office (Coordinating Investigator)
Locations (18):
- United States (18):
  - HonorHealth Research Institute, Scottsdale, Arizona
  - University of California Los Angeles, Los Angeles, California
  - Pacific Hematology Oncology Associates, San Francisco, California
  - The Angeles Clinic and Research Institute - West Los Angeles Office, Santa Monica, California
  - University of California Los Angeles, Santa Monica, California
  - Florida Cancer Specialists, Sarasota, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - The University of Chicago, Chicago, Illinois
  - Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Washington University School of Medicine Siteman Cancer Center, St Louis, Missouri
  - John Theurer Cancer Center, Hackensack, New Jersey
  - New York University Medical Oncology Associates, New York, New York
  - Weill Cornell Medicine, New York, New York
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - The Miriam Hospital, Providence, Rhode Island
  - Baylor Scott and White Center for Advanced Heart and Lung Disese, Dallas, Texas
  - Huntsman Cancer Institute and Hospital, Salt Lake City, Utah
  - Swedish Medical Oncology - First Hill, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Up to 111 evaluable patients were to be enrolled: 42 patients with melanoma, 42 patients with gastric/gastroesophageal junction (GEJ) adenocarcinoma, and 27 patients with CRC-MSS.
Groups:
- VE800 combination treatment with nivolumab: Subjects received 5 days of oral vancomycin, followed by daily VE800 in combination with nivolumab every 4 weeks.
  VE800: VE800 is a PO LBP consisting of 11 distinct nonpathogenic, nontoxigenic, commensal bacterial strains manufactured under GMP conditions. These strains were selected for their ability to induce an immune response.
  Nivolumab: Nivolumab is an approved medication that blocks antibodies for certain types of cancer.
  Vancomycin Oral Capsule: Vancomycin is an antibiotic used to treat or prevent infection.
Period: Overall Study
Arm/Group | VE800 combination treatment with nivolumab
Started | 56
gastric/GEJ adenocarcinoma | 20
Melanoma | 20
CRC-MSS | 14
not treated with VE800 | 2
Completed | 0
Not Completed | 56

BASELINE CHARACTERISTICS:
Population: Excludes one subject with gastric/GEJ adenocarcinoma who discontinued before beginning pretreatment.
Arm/Group | VE800 combination treatment with nivolumab
Number analyzed (Participants) | 55
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Analyzed separately for each tumor type.
  years
    Melanoma: number analyzed (Participants) | 21
    Melanoma | 60.2 (17.53)
    Gastric/GEJ: number analyzed (Participants) | 20
    Gastric/GEJ | 62.6 (11.51)
    CRC-MSS: number analyzed (Participants) | 14
    CRC-MSS | 56.6 (13.44)
    Total | 60.1 (14.47)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Two of the 56 enrolled subjects did not receive VE800/nivolumab. One subject in the melanoma group received vancomycin only and is included in the baseline characteristics analysis; one subject in the gastric/GEJ adenocarcinoma group did not receive any study-related treatment and is not included in this analysis.
  Participants
    Melanoma: number analyzed (Participants) | 21
    Melanoma: Female | 11
    Melanoma: Male | 10
    Gastric/GEJ: number analyzed (Participants) | 20
    Gastric/GEJ: Female | 7
    Gastric/GEJ: Male | 13
    CRC-MSS: number analyzed (Participants) | 14
    CRC-MSS: Female | 6
    CRC-MSS: Male | 8
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Two of the 56 enrolled subjects did not receive VE800/nivolumab. One subject in the melanoma group received vancomycin only and is included in the baseline characteristics analysis; one subject in the gastric/GEJ adenocarcinoma group did not receive any study-related treatment and is not included in this analysis.
  Participants
    Melanoma: number analyzed (Participants) | 21
    Melanoma: American Indian or Alaska Native | 0
    Melanoma: Asian | 0
    Melanoma: Native Hawaiian or Other Pacific Islander | 0
    Melanoma: Black or African American | 0
    Melanoma: White | 21
    Melanoma: More than one race | 0
    Melanoma: Unknown or Not Reported | 0
    Gastric/GEJ: number analyzed (Participants) | 20
    Gastric/GEJ: American Indian or Alaska Native | 0
    Gastric/GEJ: Asian | 1
    Gastric/GEJ: Native Hawaiian or Other Pacific Islander | 0
    Gastric/GEJ: Black or African American | 1
    Gastric/GEJ: White | 17
    Gastric/GEJ: More than one race | 0
    Gastric/GEJ: Unknown or Not Reported | 1
    CRS/MSS: number analyzed (Participants) | 14
    CRS/MSS: American Indian or Alaska Native | 0
    CRS/MSS: Asian | 0
    CRS/MSS: Native Hawaiian or Other Pacific Islander | 0
    CRS/MSS: Black or African American | 1
    CRS/MSS: White | 13
    CRS/MSS: More than one race | 0
    CRS/MSS: Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability of VE800 in Combination With Nivolumab: Number of Participants With Adverse Events
Description: Safety and tolerability of VE800 in combination with nivolumab: Number of Participants with Adverse Events
Time Frame: From the first dose to the last dose (up to 56.7 weeks), plus 100 days of post-treatment follow-up
Population: The analysis population included all subjects who received at least one dose of VE800 or nivolumab. Total number of subjects with at least 1 Treatment Emergent Adverse Event Reported
Measure: Number; unit: participants
Groups:
- VE800 combination treatment with nivolumab (Melanoma); VE800 combination treatment with nivolumab (Gastric); VE800 combination treatment with nivolumab (Colorectal); VE800 combination treatment with nivolumab (Total): Subjects received 5 days of oral vancomycin, followed by daily VE800 in combination with nivolumab every 4 weeks.
  VE800: VE800 is a PO LBP consisting of 11 distinct nonpathogenic, nontoxigenic, commensal bacterial strains manufactured under GMP conditions. These strains were selected for their ability to induce an immune response.
  Nivolumab: Nivolumab is an approved medication that blocks antibodies for certain types of cancer.
  Vancomycin Oral Capsule: Vancomycin is an antibiotic used to treat or prevent infection.
Arm/Group | VE800 combination treatment with nivolumab (Melanoma) | VE800 combination treatment with nivolumab (Gastric) | VE800 combination treatment with nivolumab (Colorectal) | VE800 combination treatment with nivolumab (Total)
Number analyzed (Participants) | 20 | 20 | 14 | 54
participants
  Any Treatment-emergent Adverse Event | 16 | 19 | 12 | 47
  Any Treatment Related Adverse Event | 9 | 9 | 6 | 24
  Treatment Related Adverse Event : Vancomycin Related | 1 | 3 | 1 | 5
  Treatment Related Adverse Event : Nivolumab Related | 8 | 8 | 5 | 21
  Treatment Related Adverse Event : VE800 Related | 3 | 3 | 3 | 9
  Any Grade 3 or Greater Adverse Event | 6 | 8 | 2 | 16
  Grade 3 or Greater Adverse Event : Vancomycin Related | 0 | 1 | 0 | 1
  Grade 3 or Greater Adverse Event: Nivolumab Related | 0 | 3 | 0 | 3
  Grade 3 or Greater Adverse Event: VE800 Related | 0 | 1 | 0 | 1
  Any Serious Adverse Event | 5 | 9 | 2 | 16
  Serious Adverse Event: Vancomycin Related | 0 | 0 | 0 | 0
  Serious Adverse Event: Nivolumab Related | 0 | 3 | 1 | 4
  Serious Adverse Event: VE800 Related | 0 | 1 | 0 | 1
  Any Adverse Events of Special Interest | 1 | 2 | 0 | 3
  Adverse Events of Special Interest: Vancomycin Related | 0 | 0 | 0 | 0
  Adverse Events of Special Interest: Nivolumab Related | 1 | 2 | 0 | 3
  Adverse Events of Special Interest: VE800 Related | 1 | 1 | 0 | 2
  Any Immune-Related Adverse Events | 1 | 2 | 0 | 3
  Immune-Related Adverse Events: Vancomycin Related | 0 | 0 | 0 | 0
  Immune-Related Adverse Events: Nivolumab Related | 1 | 2 | 0 | 3
  Immune-Related Adverse Events: VE800 Related | 1 | 0 | 0 | 1
  Any Adverse Events Leading to Discontinuation of any Study Drug | 1 | 1 | 0 | 2
  Adverse Events Leading to Discontinuation of any Study Drug: Vancomycin Related | NA — Not a study drug. | NA — Not a study drug. | NA — Not a study drug. | NA — Not a study drug.
  Adverse Events Leading to Discontinuation of any Study Drug: Nivolumab Related | 0 | 1 | 0 | 1
  Adverse Events Leading to Discontinuation of any Study Drug: VE800 Related | 0 | 1 | 0 | 1
  Any Adverse Events Leading to Interruption of Study Drug | 0 | 5 | 3 | 8
  Adverse Events Leading to Interruption of Study Drug: Vancomycin Related | NA — Not a study drug. | NA — Not a study drug. | NA — Not a study drug. | NA — Not a study drug.
  Adverse Events Leading to Interruption of Study Drug: Nivolumab Related | 0 | 2 | 3 | 5
  Adverse Events Leading to Interruption of Study Drug: VE800 Related | 0 | 0 | 0 | 0
  Any Adverse Events Leading to Study Discontinuation | 0 | 1 | 0 | 1
  Adverse Events Leading to Study Discontinuation: Vancomycin Related | 0 | 0 | 0 | 0
  Adverse Events Leading to Study Discontinuation: Nivolumab Related | 0 | 1 | 0 | 1
  Adverse Events Leading to Study Discontinuation: VE800 Related | 0 | 1 | 0 | 1
  Any Adverse Event with an Outcome of Death | 0 | 0 | 0 | 0

2. Primary Outcome: Objective Response Rate (ORR)
Description: Objective Response Rate (ORR) Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: 18 months (first patient enrolled to last patient visit completed)
Population: The analysis population included all subjects who received at least one dose of VE800 or nivolumab.
Measure: Count of Participants; unit: Participants
Arm/Group | VE800 combination treatment with nivolumab
Number analyzed (Participants) | 54
Participants
  Gastric: number analyzed (Participants) | 20
  Gastric | 1
  Melanoma: number analyzed (Participants) | 20
  Melanoma | 0
  CRC: number analyzed (Participants) | 14
  CRC | 0

3. Secondary Outcome: Duration of Response (DOR)
Description: Defined as the time from first documentation of complete response (CR) or partial response (PR) until the time of first documentation of progressive disease (PD) according to RECIST 1.1.
  Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: Up to two years
Population: The analysis population includes all subjects who received at least one dose of VE800 or nivolumab and had an objective response.
Measure: Number; unit: months
Arm/Group | VE800 combination treatment with nivolumab
Number analyzed (Participants) | 1
months
  Gastric | 5.6
  Melanoma: number analyzed (Participants) | 0
  Colorectal: number analyzed (Participants) | 0

4. Secondary Outcome: Best Overall Response
Description: Best response among all overall responses from cycle 1 day 1 (C1D1) until disease progression or start of new anticancer therapy.
  Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: Up to 2 years
Population: The analysis population included all subjects who received at least one dose of VE800 or nivolumab.
Measure: Count of Participants; unit: Participants
Arm/Group | VE800 combination treatment with nivolumab
Number analyzed (Participants) | 54
Participants
  CRC: number analyzed (Participants) | 14
  CRC: CR | 0
  CRC: NE | 0
  CRC: Unknown | 1
  CRC: PR | 0
  CRC: SD | 3
  CRC: PD | 10
  Melanoma: number analyzed (Participants) | 20
  Melanoma: CR | 0
  Melanoma: Unknown | 2
  Melanoma: PR | 0
  Melanoma: NE | 0
  Melanoma: SD | 9
  Melanoma: PD | 9
  Gastric: number analyzed (Participants) | 20
  Gastric: CR | 0
  Gastric: NE | 0
  Gastric: Unknown | 1
  Gastric: SD | 2
  Gastric: PD | 16
  Gastric: PR | 1

5. Secondary Outcome: Disease Control Rate (DCR)
Description: The percentage of patients who have achieved complete response (CR), partial response (PR), or stable disease (SD) from cycle 1 day 1 (C1D1) until disease progression (DP) or start of new anticancer therapy.
  Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: Up to 2 years
Population: The analysis population included all subjects who received at least one dose of VE800 or nivolumab.
Measure: Count of Participants; unit: Participants
Arm/Group | VE800 combination treatment with nivolumab
Number analyzed (Participants) | 54
Participants
  Gastric: number analyzed (Participants) | 20
  Gastric | 3
  Melanoma: number analyzed (Participants) | 20
  Melanoma | 9
  CRC: number analyzed (Participants) | 14
  CRC | 3

6. Secondary Outcome: Progression-Free Survival (PFS)
Description: Progression-Free Survival (PFS) is defined as the time from start of treatment to the earlier date of assessment of progression or death by any cause in the absence of progression.
  Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: From the first dose to the last dose (up to 56.7 weeks), plus 100 days of post-treatment follow-up and then follow-up for survival every 90 days.
Population: The analysis population included all subjects who received at least one dose of VE800 or nivolumab.
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | VE800 combination treatment with nivolumab
Number analyzed (Participants) | 54
months
  Gastric: number analyzed (Participants) | 20
  Gastric | 1.8 [1.7 to 1.8]
  Melanoma: number analyzed (Participants) | 20
  Melanoma | 1.9 [1.8 to 3.7]
  CRC: number analyzed (Participants) | 14
  CRC | 1.8 [1.7 to 2.1]
  Total | 1.8 [1.8 to 1.9]

7. Secondary Outcome: Overall Survival (OS)
Description: Overall Survival (OS) as measured from the date of start of treatment to the date of death by any cause will also be evaluated.
Time Frame: 18 months (first patient enrolled to last patient visit completed)
Population: The analysis population included all subjects who received at least one dose of VE800 or nivolumab.
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | VE800 combination treatment with nivolumab
Number analyzed (Participants) | 54
months
  Gastric: number analyzed (Participants) | 20
  Gastric | 5.8 [4.2 to 11.0]
  Melanoma: number analyzed (Participants) | 20
  Melanoma | NA [lower limit 6.5] — The point estimate of median/quartiles by Brookmeyer and Crowley is not located exactly in the middle of the confidence interval. The upper bound of CI is missing due to sparseness of the data, meaning that there are few data points, few events occurring, or a large number of ties.
  Colorectal: number analyzed (Participants) | 14
  Colorectal | 7.6 [lower limit 5.0] — The point estimate of median/quartiles by Brookmeyer and Crowley is not located exactly in the middle of the confidence interval. The upper bound of CI is missing due to sparseness of the data, meaning that there are few data points, few events occurring, or a large number of ties.

8. Secondary Outcome: Detection of VE800 Bacterial Strain Colonization in Stool
Description: Detection of VE800 bacterial strain colonization in stool was measured by pharmacokinetics (PK) of VE800
Time Frame: 18 months (first patient enrolled to last patient visit completed)
Reporting Status: Not Posted

9. Secondary Outcome: Degree of VE800 Bacterial Strain Colonization in Stool
Description: Measured by pharmacokinetics (PK) of VE800 colonization in stool
Time Frame: 18 months (first patient enrolled to last patient visit completed)
Reporting Status: Not Posted

10. Secondary Outcome: Duration of VE800 Bacterial Strain Colonization in Stool
Description: Measured by pharmacokinetics (PK) of VE800 colonization in stool
Time Frame: 18 months (first patient enrolled to last patient visit completed)
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: From the first dose to the last dose (up to 2 years), plus 100 days of post-treatment follow-up.
Description: AEs were recorded from the day of signing the ICF until 100 days after the last dose of study treatment or until alternate anticancer therapy was initiated, whichever occurred first. Thereafter, only SAEs were recorded during survival follow-up period or until alternate anticancer therapy was initiated. SAEs occurring after the start of a new treatment were reported if considered to be related to study treatment by the investigator.
Arm/Group | VE800 combination treatment with nivolumab (Melanoma) | VE800 combination treatment with nivolumab (Gastric) | VE800 combination treatment with nivolumab (Colorectal) | VE800 combination treatment with nivolumab (Total)
All-Cause Mortality (participants affected / at risk) | 9/21 | 12/21 | 10/14 | 31/56
Serious Adverse Events (participants affected / at risk) | 5/21 | 9/21 | 2/14 | 16/56
Other Adverse Events (participants affected / at risk) | 13/21 | 16/21 | 11/14 | 40/56
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | VE800 combination treatment with nivolumab (Melanoma) (N=21) | VE800 combination treatment with nivolumab (Gastric) (N=21) | VE800 combination treatment with nivolumab (Colorectal) (N=14) | VE800 combination treatment with nivolumab (Total) (N=56)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 2
Plural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 2
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 2 | 0 | 2
Abdominal Pain (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Gastrointestinal Fistula (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Intestinal Perforation (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Arthritis Infective (Infections and infestations) | 1 | 0 | 0 | 1
Bacteremia (Infections and infestations) | 1 | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 1 | 0 | 1
Alanine aminotransferase Increased (Investigations) | 0 | 1 | 0 | 1
Aspartate Aminotransferase Increased (Investigations) | 0 | 1 | 0 | 1
Blood Creatine Phosphokinase Increased (Investigations) | 0 | 1 | 0 | 1
Troponin Increased (Investigations) | 0 | 1 | 0 | 1
Pain (General disorders) | 1 | 0 | 0 | 1
Hepatitis (Hepatobiliary disorders) | 0 | 1 | 0 | 1
Spinal Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Malnutrition (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Cancer Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Cerebrovascular Accident (Nervous system disorders) | 0 | 1 | 0 | 1
Depression (Psychiatric disorders) | 1 | 0 | 0 | 1
Superior Vena cava Syndrome (Vascular disorders) | 0 | 1 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | VE800 combination treatment with nivolumab (Melanoma) (N=21) | VE800 combination treatment with nivolumab (Gastric) (N=21) | VE800 combination treatment with nivolumab (Colorectal) (N=14) | VE800 combination treatment with nivolumab (Total) (N=56)
Diarrhea (Gastrointestinal disorders) | 6 | 3 | 4 | 13
Decreased Appetite (Metabolism and nutrition disorders) | 1 | 6 | 3 | 10
Fatigue (General disorders) | 5 | 5 | 3 | 13
Anaemia (Blood and lymphatic system disorders) | 5 | 2 | 2 | 9
Nausea (Gastrointestinal disorders) | 1 | 6 | 1 | 8
Constipation (Gastrointestinal disorders) | 2 | 4 | 1 | 7
Abdominal Pain (Gastrointestinal disorders) | 0 | 2 | 4 | 6
Vomiting (Gastrointestinal disorders) | 0 | 6 | 0 | 6
Abdominal Distention (Gastrointestinal disorders) | 0 | 2 | 1 | 3
Abdominal Pain - Upper (Gastrointestinal disorders) | 0 | 2 | 1 | 3
Dyspepsia (Gastrointestinal disorders) | 1 | 1 | 1 | 3
Dysphagia (Gastrointestinal disorders) | 0 | 3 | 0 | 3
Hyponatremia (Metabolism and nutrition disorders) | 4 | 1 | 1 | 6
Dehydration (Metabolism and nutrition disorders) | 1 | 3 | 1 | 5
Hypokalemia (Metabolism and nutrition disorders) | 1 | 3 | 0 | 4
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 | 0 | 1 | 3
Oedema Peripheral (General disorders) | 1 | 1 | 1 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 3 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 3
Plural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 3
Rash (Skin and subcutaneous tissue disorders) | 3 | 1 | 1 | 5
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 1 | 1 | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1 | 4
Urinary Tract Infection (Infections and infestations) | 1 | 2 | 0 | 3
Lymphocyte Count Decrease (Investigations) | 3 | 0 | 0 | 3
Headache (Nervous system disorders) | 2 | 0 | 1 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2019-12-11): https://cdn.clinicaltrials.gov/large-docs/58/NCT04208958/Prot_001.pdf
  • Statistical Analysis Plan (2021-03-03): https://cdn.clinicaltrials.gov/large-docs/58/NCT04208958/SAP_002.pdf